CLINICAL TRIAL: NCT05074277
Title: Skeletal Response to Simulated Night Shift (SPOTLIGHT Study)
Brief Title: Skeletal Response to Simulated Night Shift
Acronym: SPOTLIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20-3013; R01HL151332 (NIH)
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Osteoporosis; Circadian Rhythm Sleep Disorder, Shift Work Type
MeSH Terms: conditions — Osteoporosis; Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (8 hours nocturnal sleep) (No Intervention): Inpatient protocol involves 8-hour sleep opportunity during the biological night throughout.
- Simulated Night Shift Work (Experimental): Two inpatient stays, each involving a baseline night, followed by a 3-hour afternoon nap opportunity, and then three 12-hour night shifts, with 8-hour daytime sleep opportunity in between.
  Interventions: Behavioral: Simulated short term night shift work schedule

INTERVENTIONS:
Behavioral: Simulated short term night shift work schedule — Participant sleep schedules (in the experimental arm) will be modified to simulate short-term (3 consecutive nights) night shift work schedule (kept awake at night and offered sleep opportunities during the day instead) in each of two inpatient stays.
  Arms: Simulated Night Shift Work

SUMMARY:
This small intervention study will determine if simulated short-term night shift work (NSW) negatively alters bone metabolism. The specific aim of the study is to determine if NSW acutely uncouples bone turnover markers (BTMs), if sympathetic tone is a mechanism for this disruption and if a resumption of a normal sleep/wake pattern reverses BTM uncoupling. Our hypothesis is that NSW will reversibly uncouple BTMs via increased sympathetic nervous system (SNS) tone.

ELIGIBILITY:
Inclusion Criteria

* Healthy, nonpregnant adults 20-40 years old who habitually sleep 7-9 hours during the biological night

  o Women must be premenopausal, on continuous combination oral contraception and not breastfeeding.
* Willing and able to complete a sleep diary, wear a wrist actigraphy monitor and complete a 3-6 week research study including two 4-night inpatient stays.
* Fully vaccinated against SARS-CoV-2, and willing to produce a negative COVID test result before their first inpatient stay.

Exclusion Criteria

* Regularly go to sleep after midnight.
* Night shift work within 1 year prior to study.
* Travel > 1 time zone within 4 weeks prior to the study or need to travel >1 time zone during study.
* Physical activity level/regimen incompatible with inpatient CTRC stay.
* Current smokers (or within the previous year of study)
* Positive drug test at screening or inpatient admission
* BMI > 30 kg/m2
* Individuals who are concurrently participating in another research protocol that would influence their safe participation in this study. For example, participants involved in a study that requires blood draws or ingestion of experimental medication as this would increase the risk of participation in our study and/or compromise study results.
* Any clinically significant unstable medical or surgical condition within the last year (treated or untreated), including history of a clinically significant abnormality of the neurological system (including cognitive disorders or significant head injury) or any history of seizure (including febrile seizure-sleep loss has been used clinically to induce seizures in patients with epilepsy). Given the wide range of illnesses that are encountered in medical practice, it would not be possible to provide a comprehensive list of each and every disease that could serve as grounds for exclusion for the subject. However, the following is a list of illness categories that would certainly be grounds for exclusion: Connective Tissue and Joint Disorders; Neurologic/cognitive Disorders; Musculoskeletal Disorders; Immune Disorders; Chronobiologic Disorders; Cardiovascular Disorders; Respiratory Disorders; Kidney Disorders; Infectious Diseases; Hematopoietic Disorders; Neoplastic Diseases; and Endocrine and Metabolic Diseases.
* Self-reported or newly diagnosed medical condition that is still being investigated or is not under good control, including those identified on screening labs such as:

  o Out-of-range values measured on a fasting blood sample: glucose > 100 mg/dl, thyroid stimulating hormone <0.5 or >5.0 uU/ml, abnormal alkaline phosphatase <39 or >117 U/l, creatinine, or hemoglobin <14.5 g/dl men
* Any clinically significant psychiatric condition, as defined by DSM-V. Individuals with a history of most psychiatric illnesses or psychiatric disorders will be excluded, such as but not limited to depression, anxiety, alcoholism, drug dependency, schizophrenic disorders, and personality disorders (performed by medical history and physician interview). However, a personal history of limited prior counseling, psychotherapy (e.g., for adjustment reactions) will NOT be exclusionary.
* Evaluation of Psychiatric/Psychological Suitability:

  * Inability to demonstrate a full understanding of the requirements and demands of the study.
  * Each participant will complete psychological screening questionnaires. Exclusionary: Center for Epidemiological Studies Depression (CES-D) > 16. Subject responses to the CES-D are reviewed immediately and appropriate referrals are made if necessary.
  * Individuals who are unaware of specific psychiatric diagnoses who have a history of having been treated with antidepressants, neuroleptic medications or major tranquilizers will be excluded from study.
  * Use of anti-depressants or any like therapeutics prescribed by a physician is exclusionary
* Individuals with any clinically significant sleep disorder; Diagnosis or symptoms of sleep disorders (history of significant parasomnia as an adult [night terrors, frequent sleep walking], insomnia, including but not limited to hypersomnias such as apnea, periodic limb movements, narcolepsy). Sleep disorders will be screened by self-report and physician interview including use of validated sleep questionnaires (PSQI, Epworth sleepiness scale, and Berlin sleep questionnaire for sleep apnea). The following scores will be used to exclude those with sleep disorders: PSQI >5, Epworth Sleepiness Scale >9.
* Individuals on medications known to affect bone turnover (e.g., glucocorticoids, osteoporosis medications);
* Use of medications/supplements/drugs that impact sleep or bone metabolism (such as but not limited to sleep medications, marijuana, etc.) within one month (participants can be studied at a later date).
* Dwelling below Denver altitude (1,600 m) 1 month prior to enrollment.
* Greater than moderate caffeine (>500 mg/day) or alcohol use (>14 standard drinks/ week or >5 drinks in one sitting)
* Inability to travel to the CU-AMC campus for study visits.
* Individuals with restrictive diets (e.g., vegan)
* Individuals with 25OHD < 20 ng/mL (may be studied at a later date)
* Individuals with eGFR < 60 mL/min/1.73m2 as this is known to affect CTX measurements.
* Z-score < -2.0 for bone mineral density at the L-spine, femoral neck, or total hip on baseline DXA as compared to the DXA machine's normative database.
* Symptoms of active illness (e.g., fever) at time of enrollment; note - participant may be studied at a later date.
* Restrictive diets that cannot be accommodated by the CTRC Nutrition Core
* Any other reason that participant may not be able to safely complete the entire study, at PI discretion

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2025-12-18 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Difference in change in propeptide of type 1 procollagen (P1NP) | Baseline to day 11
  Difference in change in propeptide of type 1 procollagen (P1NP, a bone formation marker) from baseline to day 11 between the control and simulated NSW groups.

SECONDARY OUTCOMES:
Between-group differences in the change in osteocalcin. | Baseline to day 11
  Between-group differences in the change in another bone formation marker (osteocalcin)
Between-group differences in the change in CTX (C-telopeptide of type I collagen) | Baseline to day 11
  Between-group differences in the change in bone resorption marker (CTX)

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Swanson, MD, MCR, Principal Investigator — CU Anschutz
Locations (1):
- CU Anschutz, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No